CLINICAL TRIAL: NCT05727631
Title: The Effect of Mother's Gentle Human Touch Method on Preterm Pain and Mother's Anxiety Level During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, DERYA KILINÇ, PhD, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 190
Record Dates: First submitted 2022-12-12; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Venipuncture; Pain
Keywords: NEWBORN; PRETERM; GENTLE HUMAN TOUCH; PAİN
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Intervention Model Description: Preterm babies who apply to the blood collection room to draw blood, will be included in the experimental and control group. Randomization was done at www.randomizer.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gentle human touch (Experimental): In the study, after the mother in the experimental group was dressed in a clean apron, she was allowed to wash and disinfect her hands. When the temperature of the mother's hand was measured with a non-contact thermometer, it was allowed to warm it under a radiant heater until it reached 34 ºC. The mother, who was informed about the method before, was allowed to place the palm of one hand on the baby's crown, with her fingertips touching the eyebrow line. She placed her other hand on her lower abdomen, encircling the baby's waist and hips. It has been provided to perform sensitive touch operation without pressure and massage. The mother started the gentle touch method 5 minutes before the blood draw, and continued to do the touching during the blood draw and 5 minutes after the blood draw was finished.
  Interventions: Other: gentle human touch
- Control group (No Intervention): The standard procedure of the clinic was applied to preterm infants in the control group. In the standard procedure of the clinic, the mother was with her baby in the blood collection room and did not perform any procedure.
  IN ALL BABIES IN THE CONTROL AND EXPERIMENTAL GROUP., Before the procedure, 5 minutes after the procedure and 20 minutes after the procedure, the mother filled out the STAI-I form. The NIPS scale to measure the infant's pain was scored by two independent observers before, during, and five minutes after the procedure. KTA, SPO2 values of the baby were recorded before, during and five minutes after the procedure. The baby's crying time was started when the crying started, and stopped when the crying stopped.

INTERVENTIONS:
Other: gentle human touch — Mother will apply gentle human touch touch technique during venous blood collection from preterm babies between 32-37 weeks of gestation
  Other Names: yok
  Arms: gentle human touch

SUMMARY:
Newborns are frequently exposed to acute or chronic pain experience due to different invasive interventions. The American Academy of Pediatrics (AAP) recommends minimizing the pain associated with invasive procedures. Reduction of pain primarily requires accurate assessment of pain, and treatment with pharmacological/nonpharmacological interventions.

Touch is one of the first senses developed in the newborn. Gentle Human Touch (Gentle Human Touch) is one of the therapeutic touch methods. Gentle touch, which is a simple and applicable method in newborns, is a non-invasive touch technique that does not require special equipment and technology. The gentle touch method is a sensitive tactile stimulation applied to the skin, without stroking or massage, and provides a relaxing effect on the baby. Studies have shown that the gentle touch method increases the sleep level of preterm infants, reduces pain, stress and cortisone levels, reduces restlessness and keeps the heart rate under control.

Newborns need their parents, especially their mothers, to be by their side during any kind of intervention. For this reason, the presence of the parent next to the newborn during invasive procedures and the primary role in nonpharmacological interventions provides optimal comfort for the nurse, the newborn and the caregiver. When using nonpharmacological methods, it is important to take advantage of the family-centered care model. Family-centered care is a model of care based on cooperation between health professionals and children's families in the planning, delivery and evaluation of health Decency. Its general objective is to improve the quality of health services for children and families, to increase the satisfaction of families and health professionals, and to ensure the effective use of personnel.

Accordingly, this thesis study was planned in a randomized controlled experimental design type in order to determine the importance of family-centered care model and parents' participation in the procedures and the effect of gentle touch method applied by mothers during bloodletting on preterm pain level, physiological parameters, crying time and anxiety level of the mother.

DETAILED DESCRIPTION:
June December 2021-Dec 2021, the universe of the research will consist of preterm infants and mothers admitted to Istanbul Zeynep Kamil Women and Children's Diseases Training and Research Hospital Neonatal Outpatient Clinic. The sample will be composed of mothers and preterm infants who have undergone bloodletting between these dates, who meet the sample selection criteria, and who volunteer to participate in the study Dec. At the beginning of the data collection phase, power analysis will be performed to determine the number of samples. Groups of babies will be determined using simple randomization method in computer environment.

Data Collection Process After obtaining the permissions of the ethics committee and the institution of the research, the subject and purpose of the research will be explained to all medical personnel working in the neonatal outpatient clinic of the hospital where the research will be conducted, and the methods to be applied in the research will be explained. After the parents of the babies who meet the case selection criteria are informed about the research, their oral and written consents will be obtained through the "Informed Consent Form". It will be determined by computerized simple randomization method which mothers and their babies who are willing to participate in the research and who meet the sample selection criteria will be included in which group (www.randomizer.org ). The experimental group and the control group will be fitted with a pulse oximeter device 5 minutes before the start of the blood collection procedure and it will be ensured that it is attached until 5 minutes after the procedure. 5 Minutes before the procedure, the procedure sequence and 5 minutes after the procedure, the baby's pain score, the number of heart beats, the oxygen saturation value and the mother's anxiety level will be recorded. The crying time will be recorded as the time elapsed from the moment the baby starts crying until the crying ends. All measurements will be measured by two independent observers and recorded in the observation form. The blood collection procedure will be performed by the same nurse in each of the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Between 32 and 37 gestational weeks,
* The first blood collection attempt is successful,
* Health follow-ups performed after childbirth are considered healthy by the physician,

Exclusion Criteria:

* Analgesic given up to 6 hours before the procedure,
* With a congenital anomaly, • With any disease,

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PRETERM PAİN | AT THE FIRST MINUTE OF VENİPUNCTURE
  Neonatal Infant Pain Scale
MOTHER'S ANXIETY | FIVE MINUTES AFTER VENIPUNCTURE
  State-Trait Anxiety Scale

SECONDARY OUTCOMES:
HEART RATE | AT THE FIRST MINUTE OF VENİPUNCTURE
  Measured 3 times in total
OXYGEN SATURATION | AT THE FIRST MINUTE OF VENİPUNCTURE
  Measured 3 times in total
CRYING TIME | METER STARTED WHEN BABY CRYING DURING THE PROCEDURE, STOPPED WHEN CRYING STOPPED
  measured with a stopwatch

CONTACTS AND LOCATIONS:
Overall Officials: DERYA KILINÇ, 1, Principal Investigator — ISTANBUL CERRAHPAŞA
Locations (1):
- Istanbul Provincial Health Directorate Zeynep Kamil Women and Children Diseases Traning and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdallah B, Badr LK, Hawwari M. The efficacy of massage on short and long term outcomes in preterm infants. Infant Behav Dev. 2013 Dec;36(4):662-9. doi: 10.1016/j.infbeh.2013.06.009. Epub 2013 Aug 7. PMID 23932956
- [Result] Akcan, E., & Polat, S. (2017). The role of the nurse in pain and pain management in newborns. Acıbadem University Journal of Health Sciences, (2), 64-69.
- [Result] Aydin D, Sahiner NC, Ciftci EK. Comparison of the effectiveness of three different methods in decreasing pain during venipuncture in children: ball squeezing, balloon inflating and distraction cards. J Clin Nurs. 2016 Aug;25(15-16):2328-35. doi: 10.1111/jocn.13321. Epub 2016 Apr 26. PMID 27112434
- [Result] Dur S, Caglar S, Yildiz NU, Dogan P, Guney Varal I. The effect of Yakson and Gentle Human Touch methods on pain and physiological parameters in preterm infants during heel lancing. Intensive Crit Care Nurs. 2020 Dec;61:102886. doi: 10.1016/j.iccn.2020.102886. Epub 2020 Jun 27. PMID 32601011
- [Result] Fatollahzade M, Parvizi S, Kashaki M, Haghani H, Alinejad-Naeini M. The effect of gentle human touch during endotracheal suctioning on procedural pain response in preterm infant admitted to neonatal intensive care units: a randomized controlled crossover study. J Matern Fetal Neonatal Med. 2022 Apr;35(7):1370-1376. doi: 10.1080/14767058.2020.1755649. Epub 2020 Apr 21. PMID 32316790
- [Result] Hashemi F, Taheri L, Ghodsbin F, Pishva N, Vossoughi M. Comparing the effect of swaddling and breastfeeding and their combined effect on the pain induced by BCG vaccination in infants referring to Motahari Hospital, Jahrom, 2010-2011. Appl Nurs Res. 2016 Feb;29:217-21. doi: 10.1016/j.apnr.2015.05.013. Epub 2015 May 30. PMID 26856517
- [Result] Liaw JJ, Yang L, Katherine Wang KW, Chen CM, Chang YC, Yin T. Non-nutritive sucking and facilitated tucking relieve preterm infant pain during heel-stick procedures: a prospective, randomised controlled crossover trial. Int J Nurs Stud. 2012 Mar;49(3):300-9. doi: 10.1016/j.ijnurstu.2011.09.017. Epub 2011 Oct 14. PMID 22001561
- [Result] Mayfield, A. (2019). Effects of Kangaroo Mother Care on Mother-Infant Interaction: Infant Behaviors (Doctoral dissertation, Southeast Missouri State University).
- [Result] McCarthy M, Glick R, Green J, Plummer K, Peters K, Johnsey L, Deluca C. Comfort First: an evaluation of a procedural pain management programme for children with cancer. Psychooncology. 2013 Apr;22(4):775-82. doi: 10.1002/pon.3061. Epub 2012 Mar 13. PMID 22416039
- [Result] Morrow C, Hidinger A, Wilkinson-Faulk D. Reducing neonatal pain during routine heel lance procedures. MCN Am J Matern Child Nurs. 2010 Nov-Dec;35(6):346-54; quiz 354-6. doi: 10.1097/NMC.0b013e3181f4fc53. PMID 20926970
- [Result] Yilmaz, O. E., & Gözen, D. (2019). The Importance of Family Centered Care in Pediatric Nursing and Its Value in Improving the Quality of Care. Turkiye Klinikleri Child Health and Diseases Nursing-Special Topics, 5(2), 5-11.
- [Result] Zempsky WT. Optimizing the management of peripheral venous access pain in children: evidence, impact, and implementation. Pediatrics. 2008 Nov;122 Suppl 3:S121-4. doi: 10.1542/peds.2008-1055c. No abstract available. PMID 18978004
- [Derived] Kilinc D, Caglar S. The Effect of Mother's Gentle Human Touch on Preterm Neonate's Pain and Maternal Anxiety During Venipuncture in Turkiye. Res Nurs Health. 2025 Aug;48(4):487-496. doi: 10.1002/nur.22472. Epub 2025 May 20. PMID 40392177